CLINICAL TRIAL: NCT03310138
Title: RTMS for Treatment of Pain and Craving
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 42186
Record Dates: First submitted 2017-10-10; First posted 2017-10-16 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Pain, Chronic; Pain Acute
Keywords: treatment; brain stimulation
MeSH Terms: conditions — Chronic Pain; Acute Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dorsolateral Prefrontal Cortex (Active Comparator): Intervention: Real Transcranial Magnetic Stimulation
  Real Transcranial Magnetic Stimulation will be delivered to the left dorsolateral prefrontal cortex (10Hz, 110% of resting motor threshold) using a MagVenture MagPro B60 coil.
  Interventions: Device: Real Transcranial Magnetic Stimulation
- Motor Cortex (Active Comparator): Intervention: Real Transcranial Magnetic Stimulation
  Real Transcranial Magnetic Stimulation will be delivered to the left primary motor cortex (10Hz, 80% of resting motor threshold) using a MagVenture MagPro B60 coil.
  Interventions: Device: Real Transcranial Magnetic Stimulation
- Sham stimulation (Placebo Comparator): Intervention: Sham Transcranial Magnetic Stimulation
  Sham Transcranial Magnetic Stimulation will be delivered to the prefrontal cortex (10Hz, 110% of resting motor threshold) using the integrated sham system on the MagVenture MagPro B60 coil.
  Interventions: Device: Sham Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Real Transcranial Magnetic Stimulation — Transcranial magnetic stimulation (TMS) is a minimally invasive brain stimulation technology that can focally stimulate the brain of an awake individual. A localized pulsed magnetic field transmitted through a figure-8 coil (lasting only microseconds) is able to focally stimulate the cortex by depolarizing superficial neurons, which induces electrical currents in the brain. TMS pulses that are delivered repetitively and rhythmically are referred to as repetitive TMS (rTMS). In this study TMS is being delivered with the MagVenture MagPro B60 coil.
  Other Names: TMS
  Arms: Dorsolateral Prefrontal Cortex; Motor Cortex
Device: Sham Transcranial Magnetic Stimulation — The MagVenture MagPro system has an integrated active sham that passes current through two surface electrodes placed on the skin beneath the B60 coil.
  Arms: Sham stimulation

SUMMARY:
The purpose of this study is to develop repetitive transcranial magnetic stimulation (rTMS) as a potential treatment for pain in individuals on prescription opioid medication. Repetitive TMS is a non-invasive technique that uses magnetic pulses to temporarily stimulate specific brain areas in awake people (without the need for surgery, anesthetic, or other invasive procedures). This study will test whether 10 days of rTMS over the prefrontal cortex can produce a reduction in perception of pain and the desire to use opiates. TMS has been approved by the FDA as an investigational tool as well a therapy for depression.

DETAILED DESCRIPTION:
Individuals between the ages of 18 and 65 with current (past 3 months) prescription opioid use and chronic pain are being recruited. Participants will be screened on the telephone for major inclusion/exclusion criteria. Individuals meeting inclusion criteria based on the screening assessment will be set up for an appointment in the clinic. Participants will be instructed not to use alcohol, prescription opioids, or any other drugs on the day of their appointment. All study procedures will take place at the 30 Bee Street location of the Brain Stimulation Lab (BSL). The protocol contains 1 screening visit, 10 TMS visit, and 2 follow up visits. Individuals that are eligible following the screening visit will be randomized to receive real or sham TMS.

On each TMS visit participants will undergo a single 20-minute session of 10Hz real or sham rTMS (on-time=5 secs, off-time=10 secs) at up to 110% of resting motor threshold using a MagVenture MagPro TMS machine.

Primary outcomes will be:

1. change in pain sensitivity levels in the pain assessment task and
2. change in levels of opiate craving.

The investigators will use analysis of variance models with group (real rTMS vs. sham) as the between-subjects factor and time (pre- to post-TMS) as a within-subject factor. The investigators will test the hypothesis that rTMS will result in significantly lower levels of reported pain sensitivity and craving, as compared to sham. Blind interim analyses of the data will be conducted when 50% of the sample has been accrued.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65
* currently prescribed prescription opiates for pain

Exclusion Criteria:

* documented history of seizures
* unstable chronic medical illness
* currently using any medications known to lower seizure risk
* metal above the waist
* pregnancy
* history of a negative reaction to TMS

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Thermal pain threshold | Day 1 versus Day 10
  Quantitative Sensory Testing will be used to measure each participant's thresholds for sensory detection of heat, painfulness, and tolerance. The investigators will test the hypothesis that Real TMS has a larger effect on thermal pain threshold following 10 days of TMS than sham TMS.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen A Hanlon, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The data from the primary outcome measurement will be shared via manuscripts and after study completion by request to the Principal Investigator
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available immediately after first publication of the results. This is estimated to be at the end of 2018.
Access Criteria: Interested parties should contact the Principal Investigator directly